CLINICAL TRIAL: NCT04724122
Title: Perioperative Care Capacity - an Ethiopian National Cross-sectional Survey
Brief Title: Perioperative Care in Ethiopia
Status: Completed | Type: Observational
Sponsor: Network for Perioperative Critical Care (Other)
Collaborators: Debre Berhan University (Other)
Responsible Party: Sponsor
Other Study IDs: 1.1POC
Record Dates: First submitted 2021-01-22; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Perioperative Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational / Assessment only — The results of this assessment will determine the needs for future interventions

SUMMARY:
A national cross-sectional survey of surgery and anaesthesia at Ethiopian public hospital facilities.

DETAILED DESCRIPTION:
Incorporating elements from recognized surgical and anesthesia facility assessment tools the survey assesses surgery and anaesthesia at Ethiopian public hospital facilities.

The surveys assesses infrastructure, workforce, and availability of resources across all National facilities providing surgery.

An online national cross-sectional survey, designed through a consultative process involving senior clinicians - anesthesia providers, surgeons, and obstetricians.

Elements incorporated from existing tools, including the Safe Surgery Hospital Assessment Tool, World Federation of Societies of Anaesthesiologists (WFSA) Anaesthesia Facility Assessment Tool and the Lancet Commission on Global Surgery Surgical Assessment Tool.

Survey questions grouped into themes: infrastructure, human resources, service delivery, and the availability of medications, equipment, and guidelines.

The final quantitative survey includes 77 questions, for distribution to clinicians at a convenience sample of government hospitals providing major surgical services. Private facilities are excluded.

The online survey link sent via the N4PCc collaborator network to clinicians at each site. All collaborators and clinicians are perioperative practitioners (anesthesia providers, surgeons, obstetricians, nurses) at their respective institutions. Additional facilities with no N4PCc collaborator contacted via the department of anesthesia at each institution. Telephone follow-up with non-responding hospitals to overcome barriers to completion, including assistance with data input where required.

ELIGIBILITY:
Inclusion Criteria:

Clinicians working at facilities providing perioperative care Clinicians working in surgery, anaesthesia or obstetrics These will be recruited to provide data on perioperative capacity at all facilities providing surgery nationally

Exclusion Criteria:

Clinicians working out-with perioperative care Facilities not providing surgical services

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clinicians working at facilities providing perioperative care e.g. working in surgery, anaesthesia or obstetrics, will be recruited to complete survey data pertaining to facility capacity and delivery of perioperative care. This will include infrastructure, capacity, workforce, service delivery.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Perioperative care capacity | 3 months
  Delivery of perioperative services at national level

CONTACTS AND LOCATIONS:
Locations (1):
- Debre Birhan University, Debre Berhan, Amhara, Ethiopia

IPD SHARING:
Plan to Share IPD: No
Individual facility or clinician or person data will not be available due to sensitive and confidential nature. Data will be summarised.